CLINICAL TRIAL: NCT06034132
Title: Effect of Two Different Healing Abutment Materials on Matrix Metalloproteinase-8 Level in Peri-implant Crevicular Fluid (a Randomised Clinical Trial)
Brief Title: Healing Abutment Materials on Matrix Metalloproteinase-8 Level in Peri-implant Crevicular Fluid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Implants_2022_MP8
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Other: Compoiste healing abutments
- Control group (Active Comparator)
  Interventions: Other: Stock healing abutments

INTERVENTIONS:
Other: Stock healing abutments — 2ND stage surgery will be performed and stock healing abutment were placed
  Arms: Control group
Other: Compoiste healing abutments — 2ND stage surgery will be performed and composite healing abutment were placed
  Arms: Test group

SUMMARY:
Numerous materials are nowadays used in the fabrication of healing abutments to be used for dental implants. soft tissue response to different healing abutment materials is still to be unraveled. the Aim of this study is to compare the soft tissue response to titanium stock healing abutments to customized composite healing abutments through assessing the level of matrix metalloproteinase-8 in the peri-implant crevicular fluid

ELIGIBILITY:
Inclusion Criteria:

* Patients with no systemic and/or oral health disease
* absence of any lesions in the oral cavity
* wide band of keratinized tissue more than 1mm at implant site

Exclusion Criteria:

* smoking more than 20 cigarettes per day
* localized radiation therapy of the oral cavity,
* antitumor chemotherapy, liver diseases, blood diseases, kidney diseases, immunosuppressed patients, patients taking corticosteroids, pregnancy, inflammatory and autoimmune diseases of the oral cavity

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change in MMP8 levels | at 2 weeks and 4 weeks
  Measuring MMP-8 level around composite and titanium healing abutments with ELISA kit

SECONDARY OUTCOMES:
Change in gingival condition | at 2 weeks and 4 weeks
  Modified gingival index was used to assess gingival condition The MGI uses a rating score between 0 and 4 0 = absence of inflammation
  1. = mild inflammation
  2. = mild inflammation
  3. = moderate inflmmation
  4. = severe inflammation
Change in gingival bleeding | at 2 weeks and 4 weeks
  Bleeding index will be recorded as present or absent
Change in plaque accumulation | at 2 weeks and 4 weeks
  Plaque index 0: No plaque is in the area adjacent to the gingiva. Plaque index 1: There is a plaque in the form of a thin film on the gingival margin.
  Plaque index 2: There is a visible plaque in the gingival pocket and gingival margin.
  Plaque index 3: There is a dense plaque in the gingival pocket and on the gingival margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt